CLINICAL TRIAL: NCT01729481
Title: Phase II Study to Evaluatate the Efficacy of Gemcitabine Plus Erlotinib for RASH-positive Patients With Metastatic Pancreatic Cancer and Friendly Risk Circumstances
Brief Title: Gemcitabine Plus Erlotinib in RASH-positive Patients With Metastatic Pancreatic Cancer
Acronym: ML22774
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, PD Dr. med. Volker Heinemann, Clinical Professor, Ludwig-Maximilians - University of Munich
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2011-005471-17
Record Dates: First submitted 2012-10-23; First posted 2012-11-20 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; Erlotinib Hydrochloride; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RASH positive (Experimental): Run-In-Phase during 4 weeks:
  Gemcitabine 1000 mg/m², weekly Erlotinib 100 mg, weekly
  Thereafter Treatment in patients with RASH-positve outcome after 4 weeks.
  Interventions: Drug: Gemcitabine; Drug: Erlotinib
- RASH-negative (Active Comparator): Run-In-Phase during 4 weeks:
  Gemcitabine 1000 mg/m², weekly Erlotinib 100 mg, weekly
  RASH-negative patients quit treatment with Gemcitabine + Erlotinib and continue treatment with FOLFIRINOX:
  Oxaliplatin 85mg/m2 Irinotecan 180 mg/m2 Folinic acid 400 mg/m2 5-FU 400 mg/m2 bolus iv 5-FU 2400 mg/m2 46-hours continous infusion
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: Irinotecan; Drug: 5-FU

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m² iv weekly
  Other Names: Gemzar
  Arms: RASH positive
Drug: Erlotinib — 100mg, once per day
  Other Names: Tarceva
  Arms: RASH positive
Drug: Oxaliplatin — 85mg/m², q2weeks
  Other Names: Eloxatin
  Arms: RASH-negative
Drug: Folinic Acid — 400 mg/m², q2weeks
  Other Names: Leucovorin
  Arms: RASH-negative
Drug: Irinotecan — 180 mg/m², q2weeks
  Other Names: Campto
  Arms: RASH-negative
Drug: 5-FU — 400 mg/m² Day 1; 2400 mg/m² 46 hour invusion, q2weeks
  Other Names: 5-Flourouracil
  Arms: RASH-negative

SUMMARY:
In the current study it is examined whether patients with good risk factors (age <75 years, total serum bilirubin < 1,5xULN, no history of cardiovascular diseases) treated with gemcitabine and erlotinib who developed skin rash of any grade during the first 4 weeks of treatment have a comparable outcome as patients who receive FOLFIRINOX.

DETAILED DESCRIPTION:
The study by Burris et al. 1997 revealed a superiority of gemcitabine vs. 5-FU in terms of improvement of general condition, pain symptoms and overall survival in patients with locally advanced or metastatic pancreatic cancer. Subsequently, gemcitabine was established as a standard treatment for locally advanced and metastatic pancreatic cancer.

In a series of studies gemcitabine was combined with other chemotherapeutic agents or targeted therapies. For the first time, the PA.03 study showed a significant improvement of overall survival. Patients who were treated with gemcitabine plus erlotinib had a survival of 6.24 months, compared with 5.91 months for those treated with gemcitabine plus placebo (HR 0.82, 95% CI 0.69-0.99, p=0.038). The one-year-survival rate was 23% for gemcitabine plus erlotinib vs. 17% for gemcitabine plus placebo.

In a subgroup analysis of the PA.03 study, patients developing a skin rash NCI CTC ≥ grade 2 had an advanced survival (one-year-survival rate 43%) vs. those with grade 1 or 0 (one-year-survival rate 16% and 9%, respectively). Later studies confirmed the correlation between skin rash and survival.

While patients developing a skin rash of any grade seem to profit most from treatment with erlotinib, the prognosis for those without rash is rather dismal. In this population, survival varied between 3.3 and 4.8 months in clinical trials (Verslype et al. 2009, Boeck et al. 2010, Manzano et al. 2010). In this patients, a modification of the treatment strategy should be considered. Which kind of treatment might lead to optimal results in these patients is not yet clear.

In patients with excellent general condition complying with further prerequisits (age <75 years, total serum bilirubin < 1,5xULN, no history of cardiovascular diseases) the French Prodige study-group could show a statistical superiority for the gemcitabine-free FOLFIRINOX-scheme in terms of overall survival, progression free survival and response rate compared to gemcitabine alone. However, this superiority was gained at the expense of treatment tolerability. During treatment with FOLFIRINOX a grade 3-4 neutropenia was observed in 5.4% and a grade 3-4 diarrhea in 12.7% of patients (Conroy et al. 2011). For patients who comply with the above-named criteria FOLFIRINOX is considered an established standard of care.

If a comparable efficacy of gemcitabine plus erlotinib with the published FOLFIRINOX data can be seen in the selected population, this would favour, due to the worse tolerability of FOLFIRINOX, the use of gemcitabine plus erlotinib.

In summary, the following selections are conducted during the study:

1. Selection due to the inclusion criteria for treatment with FOLFIRINOX provided by Conroy et al.
2. Selection due to the development of a skin rash within four weeks of treatment
3. No signs of clinical tumour progression within the run-in phase within the first four weeks of treatment

Patients who do not develope a skin rash of any grade should be treated with FOLFIRINOX. The efficacy of FOLFIRINOX in rash-negative patients has not yet been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically (not cytologically) confirmed metastatic pancreatic adenocarcinoma (stage IV according to UICC, each T, each N, M1 according to TNM)
* At least one measurable index lesion (CT or MRI) according to RECIST criteria (V 1.1)
* ECOG PS 0 and 1
* Age 18-75 years
* Serum bilirubin ≤1,5x ULN (a placed biliary tract stent without concurrent cholangitis is not considered a contraindication)
* Availability of tumour samples (no cytologic samples)
* Written informed consent by the patient for collecting blood- and tumour-samples for translational research according to study protocol
* Live expectancy of at least three months
* Written informed consent
* Negative pregnancy test in women with childbearing potential (to be performed within 7 days prior to treatment start)
* Adequate kidney-, liver- and bone-marrow function: neutrophils >= 1500/µl, platelets >= 100.000/µ, and hemoglobin >= 8g/dl, liver transaminases<= 2,5x ULN, in case of liver metastases <= 5x ULN, serum creatinine <= 1,25x ULN, creatinine clearance ≥ 30 ml/min
* Legal capacity of the patient
* Option for constant long-term follow-up

Exclusion Criteria:

* Resectable pancreatic carcinoma
* Locally advanced pancreatic cancer (non-resectable tumour without distant metastasis)
* Previous palliative chemotherapy for metastatic or locally advanced, non-resectable pancreatic cancer
* Previous palliative radiation or chemoradiation for locally advanced, non-resectable pancreatic cancer
* Radiation therapy within four weeks prior to study enrolment or radiation of indicator lesions
* Adjuvant Chemotherapy or Radiochemotherapy for pancreatic cancer ≤ 6 months prior to study ernrolment
* All previously occurred metastatic cancers or cured neoplasias diagnosed within the last 5 years before study enrolment
* Major surgery within 2 weeks before study start
* Chronic diarrhea
* Known glucuronidation-deficiency (Gilbert´s syndrome)
* Acute or subacute ileus or chronic inflammatory bowel disease
* Preexisting polyneuropathy > Grade I according to NCI-CTCAE v.4.0
* Relevant comorbidities which might impair patient eligibility or safety for study participation like active infections, hepatic, renal or metabolic diseases
* Clinically significant cardiovascular diseases within 12 months prior to study start (e.g. unstable angina pectoris, myocardial infarction, heart failure ≥ NYHA II, cardiac arrhythmias requiring treatment)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
1-year Survial rate of "good-risk" patients | Follow-Up Phase (1.5 years)
  1-year Survial rate of "good-risk" patients of patients under gemcitabine plus erlotinib with RASH

SECONDARY OUTCOMES:
Evalutation of overall response rate, disease control rate and progression free survival | Approximately 12 months
  Evaluation of Parameters by RASH positve and negative patients:
  * ORR
  * DCR
  * PFS
  * OS
Evaluation of adverse events | Treatment Phase (1.5 Years)
  Assesment with NCI-CTCAE V4.0 Evalutation of side effects including picture documentation of skin-rash
Translational Projects | Approximately 24 months
  * Evaluation of Parameters for EGFR signal transduction
  * Evaluation Molecularbiological Parametrs of RASH
  * Picture Documentation of RASH. Corellation with clinical and molecularbiological Parameters

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, Professor, Principal Investigator — Medical Department III and Comprehensive Cancer Center
Locations (1):
- University of Munich, Munich, Germany

REFERENCES:
- [Derived] Weiss L, Heinemann V, Fischer LE, Gieseler F, Hoehler T, Mayerle J, Quietzsch D, Reinacher-Schick A, Schenk M, Seipelt G, Siveke JT, Stahl M, Vehling-Kaiser U, Waldschmidt DT, Dorman K, Zhang D, Westphalen CB, von Bergwelt-Baildon M, Boeck S, Haas M. Three-month life expectancy as inclusion criterion for clinical trials in advanced pancreatic cancer: is it really a valid tool for patient selection? Clin Transl Oncol. 2024 May;26(5):1268-1272. doi: 10.1007/s12094-023-03323-1. Epub 2023 Oct 4. PMID 37794220
- [Derived] Haas M, Siveke JT, Schenk M, Lerch MM, Caca K, Freiberg-Richter J, Fischer von Weikersthal L, Kullmann F, Reinacher-Schick A, Fuchs M, Kanzler S, Kunzmann V, Ettrich TJ, Kruger S, Westphalen CB, Held S, Heinemann V, Boeck S. Efficacy of gemcitabine plus erlotinib in rash-positive patients with metastatic pancreatic cancer selected according to eligibility for FOLFIRINOX: A prospective phase II study of the 'Arbeitsgemeinschaft Internistische Onkologie'. Eur J Cancer. 2018 May;94:95-103. doi: 10.1016/j.ejca.2018.02.008. Epub 2018 Mar 20. PMID 29549862
- See also: Homepage of the PancreasCenter at LMU Munich — http://www.klinikum.uni-muenchen.de/Pankreaszentrum-Muenchen/de/startseitenmeldungen/index.html